CLINICAL TRIAL: NCT04713826
Title: Proof-of-concept, Multi-center, Randomized, Double-blind, Placebo-controlled, Two-way Crossover Study to Investigate the Effect Strength of BAY 2586116 on the Apnea-hypopnea-index After Repetitive Nasal Doses Compared to Placebo in 80 Valid Participants With Moderate to Severe Obstructive Sleep Apnea
Brief Title: A Trial to Learn More About How Well BAY2586116 Works and How Safe it is in Participants With Moderate to Severe Obstructive Sleep Apnea
Acronym: SPRAY-SMART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20849; 2020-000520-19 (EudraCT Number)
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive sleep apnea; OSA; AHI; Sleep lab; PSG
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAY2586116_Placebo (Experimental): Male or female participants aged above or equal to 18 years diagnosed with moderate to severe OSA will be allocated randomly to this intervention sequence.
  Participants will receive BAY2586116 in treatment period 1, and placebo in treatment period 2.
  Each intervention will be applied at home for 6 days (+1 optional day) followed by one in-house application for the overnight PSG (polysomnography).
  In total, each participant will receive up to a maximum of 7 single doses (8 single doses if optional day is used) of BAY2586116 and up to 7 single doses of placebo (8 single doses if optional day is used).
  Interventions: Drug: BAY2586116; Drug: Placebo
- Placebo_BAY2586116 (Experimental): Male or female participants aged above or equal to 18 years diagnosed with moderate to severe OSA will be allocated randomly to this intervention sequence.
  Participants will receive placebo in treatment period 1, and BAY2586116 in treatment period 2.
  Each intervention will be applied at home for 6 days (+1 optional day) followed by one in-house application for the overnight PSG.
  In total, each participant will receive up to a maximum of 7 single doses (8 single doses if optional day is used) of BAY2586116 and up to 7 single doses of placebo (8 single doses if optional day is used).
  Interventions: Drug: BAY2586116; Drug: Placebo

INTERVENTIONS:
Drug: BAY2586116 — 160 µg, nasal spray administration.
Drug: Placebo — Placebo matching BAY2586116, nasal spray administration.

SUMMARY:
Researchers are looking for a better way to treat people with obstructive sleep apnea (OSA). In people with OSA, the upper airways can narrow or close repetitively while sleeping. These breathing interruptions lead to reduction of oxygen in the blood or short arousals from sleep. Before a treatment can be approved for people to take, researchers do clinical trials to better understand its safety and how well it works.

In this trial, the researchers want to learn more about how well BAY2586116 works in a small number of participants with OSA. The trial will include about 160 men and women who have OSA and are at least 18 years old. Women can only be included in this trial if they are not able to have children naturally.

In this trial, the participants will take BAY2586116 and a placebo. A placebo looks like a treatment but does not have any medicine in it. All of the participants will take BAY2586116 through a nasal spray. They will also take the placebo as a nasal spray.

This will be a crossover trial. This means all the participants will take both trial treatments one after the other, but in a different order. The participants will take each treatment once a day for 7 days.

The researchers will use a measurement called the apnea-hypopnea-index (AHI) to measure the severity of the participants' OSA. The researchers will then compare the participants' AHI scores when they take BAY2586116 and when they take the placebo.

During study, the participants will visit their trial site 5 times. At these visits the doctors will take blood samples, do physical examinations and check the participants' heart health using an electrocardiogram (ECG). They will also ask the participants questions about how they are feeling and if they have any medical problems. At 3 of the visits, the participants will stay at the trial site overnight. At these visits, the doctors will calculate the number of times the participants stop breathing per hour of sleep. After treatment, the participants will have a final visit 7 days later so the doctors can check their health.

ELIGIBILITY:
Inclusion Criteria:

* A participant must be at least 18 years of age, at the time of signing the informed consent.
* Participants need to be diagnosed with OSA.
* 15 ≤ AHI ≤ 60 per hour documented by baseline PSG (evaluated by NOX software; manual overreading by site staff possible) and after ≥72 hours of stop of specific OSA therapy. (One re-testing allowed if e.g. sleep time is less than 4 hours or e.g. due to technical problems with PSG measurement).
* Male and/or female with non-childbearing potential. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

  * Male participants: Men of reproductive potential must agree to use at least two adequate contraception methods when sexually active.
  * Female participants: Female participants must be of non-childbearing potential, i.e. post-menopausal (no menses for at least 1 year) or surgically sterile (tubal ligation, hysterectomy, bilateral salpingectomy or bilateral oophorectomy).
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
* Ability to understand and follow study-related instructions.
* Informed consent must be signed before any study specific tests or procedures are done.

Exclusion Criteria:

* Not predominantly OSA evidenced at baseline, as judged by the investigator.
* Severely impaired breathing within two days prior to randomization (e.g. acute nasal congestion during upper airway infection).
* Participant with known allergies or hypersensitivities to the study interventions (active substances or excipients of the preparations). Known severe respiratory tract allergies e.g. allergic asthma.
* Suspected or proven active SARS-CoV-2 infection, as judged by the investigator
* Subjects with a clinical diagnosis of chronic heart failure with New York Heart Association (NYHA) class III - IV as judged by the investigator at screening visit.
* Uncontrolled arterial hypertension with diastolic blood pressure (DBP) >110 mmHg or systolic blood pressure (SBP) >180 mmHg at screening visit.
* Chronic obstructive pulmonary disease (COPD) with more than one exacerbation during the last 12 months prior to screening visit.
* Previous assignment to a study intervention during this study.
* Participation in another trial with an investigational drug within 30 days or 5 half-lives of the investigational drug, whichever is longer before first application of study intervention or concomitant participation in another clinical study with investigational medicinal product(s).
* Heavy smoking, i.e. more than 20 cigarettes or equivalent per day and/or unable to stop smoking during the stay in the sleep laboratory.
* Suspicion of drug or alcohol abuse.
* Regular daily consumption of more than 1 L of xanthine-containing beverages.
* Inability to comply with planned study procedures or to comply with study protocol requirements; this includes completing required data collection and attending required end of study/follow up study visits.
* Any other condition, which would make the participant unsuitable for this study and will not allow participation for the full planned study period (e.g. active malignancy or other condition limiting life expectancy to less than 12 months).
* Close affiliation with the investigational site; e.g. a close relative of the investigator, dependent person (e.g. employee or student of the investigational site).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Responder rates for BAY2586116 and placebo | At day -1, and day 7 in Period 1, and day 7 in Period 2
  A response is defined as reduction of apnea-hypopnea index (AHI) from baseline by ≥50%

SECONDARY OUTCOMES:
Number of participants with at least one treatment-emergent adverse event (TEAE) and maximum severity of TEAEs per participant | From first application of study intervention up to 2 days after end of treatment in each period with study intervention

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (2):
  - Ruhrlandklinik, Westdeutsches Lungenzentrum, Essen, North Rhine-Westphalia
  - Advanced Sleep Research GmbH, Berlin
- UniversitätsSpital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/